CLINICAL TRIAL: NCT03075514
Title: Ketogenic Diets as an Adjuvant Therapy in Glioblastoma: A Randomised Pilot Trial
Brief Title: Ketogenic Diets as an Adjuvant Therapy in Glioblastoma
Acronym: KEATING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liverpool (Other)
Collaborators: Walton Centre NHS Foundation Trust (Other); Vitaflo International, Ltd (Industry)
Responsible Party: Principal Investigator, Michael Jenkinson, Chief Investigator, University of Liverpool
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UoL001277
Record Dates: First submitted 2017-02-28; First posted 2017-03-09 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Glioblastoma; Glioblastoma Multiforme; Glioblastoma, Adult
Keywords: ketogenic
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Intervention Model Description: MKD and MCT ketogenic diets
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified ketogenic diet (MKD) (Active Comparator): MKD: 80% fat and 5% carbohydrate (% of total energy requirements per day).
  Interventions: Other: MKD
- Medium chain triglyceride (MCT) diet (Active Comparator): MCT: 75% fat (30% of which is medium chain fatty acids taken as a supplement) and 5% carbohydrate (% of total energy requirements per day).
  Interventions: Other: MCT

INTERVENTIONS:
Other: MKD — Modified ketogenic diet
  Arms: Modified ketogenic diet (MKD)
Other: MCT — Medium chain triglyceride ketogenic diet
  Arms: Medium chain triglyceride (MCT) diet

SUMMARY:
Glioblastoma (GB) is the commonest form of brain cancer in adults. Despite current treatment options including surgery, radiotherapy and chemotherapy, overall survival is poor. Therefore, other treatment options are being explored and there is increasing interest in the possibility of using the ketogenic diet (KD), alongside current treatment options.

The KD is a high fat, low carbohydrate diet. This encourages the body to use fat (broken down to ketones) as its primary energy source, instead of carbohydrate (broken down to glucose, a type of sugar). KDs have been considered for use in patients with GB as this type of cancer is thought to use glucose as its main energy supply, which is of short supply in this diet. Animal studies have shown KDs may make GB more responsive to radiotherapy and chemotherapy and could improve survival by slowing the cancer's growth. However, clinical studies are needed in humans to assess any possible benefits.

This trial will see patients randomly assigned to one of two types of KDs; the modified ketogenic diet (MKD) and the medium chain triglyceride ketogenic diet (MCT). Both diets follow the same high fat, low carbohydrate principles, with the MCT diet requiring the patient to take some of the fat as a supplement drink instead of as food. Patients will follow the diet for 12 weeks initially. The trial will look to enroll newly diagnosed GB patients, from The Walton Centre NHS Foundation Trust over a 12 month period.

The aim of the trial is to investigate protocol feasibility and patient impact by comparing two KDs in an NHS setting, with a view to informing future phase III clinical trials.

DETAILED DESCRIPTION:
A prospective, non-blinded, randomized, pilot study will be undertaken in patients with glioblastoma (GB). Patients will be randomized to the modified ketogenic diet (MKD) or the medium chain triglyceride ketogenic diet (MCT) for a 12 week period (primary completion). If patients wish to remain on diet, they will be offered dietetic support for a total of 12 months (secondary completion).

The trial will be open to all Walton Centre Foundation Trust patients with a newly diagnosed GB, who have undergone surgical resection or biopsy within the last four months and who are going on to receive/ are currently receiving/ have completed oncological treatments (radiotherapy or chemotherapy or chemoradiotherapy). Patients will be referred via neuro-oncology multi-disciplinary meetings and neurosurgical clinics, post histology. The diet will be offered alongside standard care, commencing within four months of surgery.

Both diets are high in fat and low in carbohydrate, but contain different types and amounts of fats. The MKD is 80% fat (predominately long chain fatty acids) and 5% carbohydrate, whilst the MCT diet is 75% fat (30% of which is medium chain fatty acids) and 10% carbohydrate.

A permuted block randomization method will be adopted, using 'sealedenvelope' randomization system. This will be set up and administered by the statistician, who is not involved with the recruiting of patients.

Patients will receive regular input from the trial dietitian. This includes clinical consultations at baseline, dietary initiation, week 6, week 12 and every 3 months thereafter and telephone consultations at weeks 1, 3 and 9. Patients will receive dietary and ketone monitoring education.

Assessments and monitoring undertaken at each consultation include anthropometry, biochemistry, compliance, tolerance, acceptability, quality of life and ketosis.

Informed consent will be obtained prior to enrollment and the patient may withdraw at any time.

An information study is also embedded into KEATING, to aid understanding of the patients' recruitment experience and viewpoints, by interviewing a sub-sample of patients and their relatives/ carers. This will enable the design of bespoke strategies to optimise recruitment to future trials related to ketogenic diets and gliomas

ELIGIBILITY:
Inclusion Criteria:

* Age ≥16 years
* Patient at The Walton Centre NHS Foundation Trust
* Performance status ≤2
* Confirmed histological diagnosis of glioblastoma
* Undergone surgical resection or biopsy and will go onto receive/ is receiving/ has received oncological treatments

Exclusion Criteria:

* Having prior use of KD
* Kidney dysfunction
* Liver dysfunction
* Gall bladder dysfunction
* Metabolic disorder
* Eating disorder
* Diabetes (requiring medication)
* Body mass index ≤ 18.5kg/m2
* Weight loss medications
* Currently pregnant or breast feeding
* Performance status ≥3

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-03-05 (Actual); Study Completion 2019-03-05 (Actual)

PRIMARY OUTCOMES:
To assess retention and drop out rates | 12 weeks
  Number of patients who start randomized treatment as a proportion of the number randomized ;
To assess retention and drop out rates | 12 weeks
  The number of patients who complete 12 weeks as a proportion of the number randomized
To assess retention and drop out rates | 12 weeks
  Description of barriers and facilitators to data collection and participant retention
To assess retention and drop out rates | 12 weeks
  The time to dietary discontinuation

SECONDARY OUTCOMES:
Estimation of recruitment rates | 12 months
  Actual recruitment compared to proposed recruitment
Enrollment of patients | 12 months
  Number of patients initiated on diet prior to starting oncological treatments.
Enrollment of patients | 12 months
  Number of patients initiated on diet during oncological treatments.
Enrollment of patients | 12 months
  Number of patients initiated on diet post oncological treatments.
Long term retention | 2 years
  Time to dietary discontinuation after week 12
Dietary adjustments required to achieve ketosis | 2 years
  Number of dietary adjustments to macronutrient composition of MCT and MKD diets required to achieve ketosis.
Self reported dietary compliance | 2 years
  Self reported by compliance rate
Calculated dietary compliance | 2 years
  Analysed by comparing macronutrient content assessed via 3 day food diaries to advised macronutrient content.
MCT compliance | 2 years
  Dose of MCT taken compared to dose advised.
Ketosis levels | 2 years
  Self reported urinary ketone levels twice daily for first 6 weeks then once per week thereafter and blood ketone and glucose levels weekly.
Dietetic time required for interventions | 2 years
  Dietetic time spent on clinical and non clinical activities relating to the trial.
Protocol refinements required | 2 years
  Number of deviations from the protocol including reasons for deviations.
Sample size estimates for future trials | 2 years
  Number of participants required for future phase III clinical trials
Quality of life | 2 years
  Change in quality of life assessed through EORTC QLQ C30 and BN 20 questionnaires
Food acceptability | 2 years
  Change in food acceptability assessed through food acceptability questionnaire
Gastrointestinal side effects | 2 years
  Number of reported gastrointestinal side effects assessed through EORTC QLQ C30 questionnaire and Common Terminology Criteria for Adverse Events.
Changes to biochemical markers | 2 years
  Changes to biochemical markers (renal, bone, LFT, lipid profiles) during the duration of the diet.
Anthropometric changes | 2 years
  Changes to anthropometry (weight, body mass index, fat mass, muscle circumference, hand grip strength) during the duration of the diet.
Completeness of data | 2 years
  Number of complete data sets for all trial outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Jenkinson, PhD, FRCS, Principal Investigator — University of Liverpool
Locations (1):
- Univeristy of Liverpool/ The Walton Centre NHS Foundation Trust, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martin-McGill KJ, Marson AG, Tudur Smith C, Jenkinson MD. Ketogenic diets as an adjuvant therapy in glioblastoma (the KEATING trial): study protocol for a randomised pilot study. Pilot Feasibility Stud. 2017 Nov 28;3:67. doi: 10.1186/s40814-017-0209-9. eCollection 2017. PMID 29209515